CLINICAL TRIAL: NCT02118467
Title: A Randomized Double Blind Trial of Vasoactive Drugs for the Management of Shock in the ICU
Brief Title: Vasoactive Drugs in Intensive Care Unit
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-0047
Record Dates: First submitted 2014-03-21; First posted 2014-04-21 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Shock
Keywords: Shock; Vasopressor agents; Norepinephrine; Epinephrine; Phenylephrine; Vasopressin; Atrial fibrillation; Tachyarrhythmia
MeSH Terms: conditions — Shock; Diabetes Insipidus; Atrial Fibrillation; Tachycardia | interventions — Norepinephrine; Epinephrine; Phenylephrine; Vasopressins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norepinephrine and epinephrine (Active Comparator): Patients will receive norepinephrine infusion per standard protocol. Dose range will be 0.03-0.3 mcg/kg/minute. Norepinephrine concentration will be 16 mg/250 mL. If a second vasopressor is required, epinephrine will be added. Dose range of epinephrine will be 0.03-0.3 mcg/kg/minute. Epinephrine concentration will be 16 mg/250 mL. The drugs norepinephrine and epinephrine will be mixed and blinded by the research pharmacy. The research pharmacist will list the dose ranges in mL/hr; this will allow the bedside nurse to program the medication per standard protocol.
  If the patient's shock is not adequately treated with the highest doses of both norepinephrine and epinephrine, additional, open-label norepinephrine will be added, and titrated to achieve target blood pressure. If the patient's shock is not adequately treated with three vasopressors, additional open-label epinephrine will be added, and titrated to achieve target blood pressure.
  Interventions: Drug: Norepinephrine; Drug: Epinephrine
- Phenylephrine and vasopressin (Active Comparator): Patients will receive phenylephrine infusion per standard protocol. Dose range will be 0.3 to 3.0 mcg/kg/minute. Phenylephrine concentration will be 160 mg/250 mL. If a second vasopressor is required, vasopressin will be added. Dose range of vasopressin will be 0.1 to 0.6 milliunits/kg/minute. Vasopressin concentration will be 40 units/250 mL. The drugs phenylephrine and vasopressin will be mixed and blinded by the research pharmacy. The research pharmacist will list the dose ranges in mL/hr; this will allow the bedside nurse to program the medication per standard protocol.
  If the patient's shock is not adequately treated with the highest doses of both phenylephrine and vasopressin, additional, open-label norepinephrine will be added, and titrated to achieve target blood pressure. If the patient's shock is not adequately treated with three vasopressors, additional open-label epinephrine will be added, and titrated to achieve target blood pressure.
  Interventions: Drug: Phenylephrine; Drug: Vasopressin

INTERVENTIONS:
Drug: Norepinephrine — Dose range 0.03 to 0.3 mcg/kg/minute, titrated to target blood pressure.
  Other Names: Levophed
  Arms: Norepinephrine and epinephrine
Drug: Epinephrine — Dose range 0.03 to 0.3 mcg/kg/minute, titrated to target blood pressure.
  Arms: Norepinephrine and epinephrine
Drug: Phenylephrine — Dose range 0.3 to 3.0 mcg/kg/minute, titrated to target blood pressure.
  Other Names: Neo-Synephrine
  Arms: Phenylephrine and vasopressin
Drug: Vasopressin — Dose range 0.1 to 0.6 milliunits/kg/minute, titrated to target blood pressure.
  Other Names: Pitressin
  Arms: Phenylephrine and vasopressin

SUMMARY:
The investigators hypothesis is that for ICU patients with shock, the use of the vasoactive drugs phenylephrine and vasopressin will reduce tachydysrhythmias when compared to norepinephrine and epinephrine. To investigate this hypothesis, the investigators are conducting a randomized double blind controlled trial comparing phenylephrine and vasopressin vs. norepinephrine and epinephrine in ICU patients with shock that is not responsive to IV fluids. All patients admitted to the adult intensive care units at the University of Chicago will be screened for eligibility.

DETAILED DESCRIPTION:
Shock, defined by inadequate tissue perfusion, is a common problem in critically ill patients. Most patients who have shock have hypotension and this is typically treated initially with intravenous fluid resuscitation in patients who are fluid responsive. If patients remain hypotensive, they are typically treated with vasoactive medications. Four of the commonly used FDA approved vasoactive medications are norepinephrine, phenylephrine, epinephrine, and vasopressin. Apart from a 2010 trial comparing norepinephrine to dopamine, there are no studies to date that have shown one of the four above-mentioned vasoactive medications to be superior to another. Accordingly, choice of vasoactive medication is based upon individual physician preference, without an outcomes-related evidence base.

Two of the four above mentioned vasoactive medications (norepinephrine and epinephrine) have chronotropic effects (i.e. the tendency to increase heart rate), while the other two (phenylephrine and vasopressin) have less of a propensity to chronotropy. The potential benefits of the chronotropic effects in patients with shock (increasing cardiac output) are offset by the potential detriments (predilection to tachydysrhythmias and myocardial ischemia).

Recent evidence suggests that tachydysrhythmias are associated with worse outcomes in ICU patients. One study demonstrated that administration of the beta blocking agent esmolol improved hemodynamic outcomes and survival in patients with septic shock. It is not clear if a vasoactive drug regimen that utilizes phenylephrine and vasopressin will be associated with lower heart rates compared to a regimen that utilizes norepinephrine and epinephrine.

The investigators hypothesis is that for ICU patients with shock, the use of the vasoactive drugs phenylephrine and vasopressin will reduce tachydysrhythmias when compared to norepinephrine and epinephrine. To investigate this hypothesis, we are conducting a randomized double blind controlled trial comparing phenylephrine and vasopressin vs. norepinephrine and epinephrine in ICU patients with shock that is not responsive to IV fluids. All patients admitted to the adult intensive care units at the University of Chicago will be screened for eligibility.

Patients will be randomized to receive either phenylephrine (0.3-3.0 mcg/kg/minute), with the addition of vasopressin (0.1-0.6 milliunits/kg/minute) if a second vasopressor is required, or norepinephrine (0.03 to 0.3 mcg/kg/minute), with the addition of epinephrine (0.03 to 0.3 mcg/kg/minute) if a second vasopressor is required. These drugs will be mixed and blinded by the research pharmacy. Only the research pharmacist will know the identity of the particular vasoactive drug. As per current standard practice, the medical team in charge of the patient will determine the target blood pressure.

In either group, if two vasoactive drugs are not adequate to raise the blood pressure to the target level, open-label norepinephrine will be added. If three vasoactive drugs are inadequate to raise the blood pressure to the target level, open-label epinephrine will be added.

There will be up to a twelve-hour period from initiation of standard, non-study vasoactive support during which the patient can be consented and enrolled. This will allow the research team to contact the patient and/or family in order to obtain informed consent. Once randomized, all patients will be initiated on study drug vasoactive support at 50 percent of the maximal infusion rate. The study drug will be titrated to maintain blood pressure and the initial non-study drug will be titrated off. The primary team will direct other aspects of patient care.

We plan to examine the following pre-specified sub-groups:

1. Patients who received corticosteroids during their ICU stay vs. patients who did not receive corticosteroids during their ICU stay
2. Patients with depressed left ventricular ejection fraction (< 40%) vs. patients with normal left ventricular ejection fraction
3. Patients with coronary artery disease vs. patients without known coronary artery disease
4. Patients with different etiologies of shock (i.e. septic, cardiogenic, hypovolemic)

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years old
2. Requirement for vasoactive drugs via a central venous catheter for the treatment of shock. Shock will be defined as mean arterial pressure less than 70 mmHg or systolic blood pressure less than 100 mmHg despite administration of at least 1000 mL of crystalloid or 500 mL of colloid, unless there is an elevation in the central venous pressure to > 12 mmHg or in the pulmonary artery occlusion pressure to > 14 mmHg coupled with signs of tissue hypoperfusion (e.g. altered mental state, mottled skin, urine output < 0.5 mL/kg body weight for one hour, or a serum lactate level of > 2 mmol per liter).

Exclusion Criteria:

1. Cardiopulmonary arrest
2. Pregnancy
3. Severe right heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 836 (Estimated)
Dates: Start 2014-05-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality | Six months

SECONDARY OUTCOMES:
Heart rate | Six months
Incidence of tachydysrhythmia | SIx months
  Including both atrial arrhythmias (i.e. atrial fibrillation, atrial flutter) as well as ventricular dysrhythmias

OTHER OUTCOMES:
Hospital length of stay | Six months
Discharge location | Six months
  i.e. to home, skilled nursing facility, nursing home, rehabilitation
ICU Complications | Six months
  Including the following:
  1. Ventilator associated pneumonia
  2. Barotrauma
  3. Gastrointestinal hemorrhage
  4. Pulmonary embolism
  5. Sacral decubitus ulcer
  6. Delirium
  7. ICU acquired weakness
ICU length of stay | Six months
Duration of mechanical ventilation | Six months
Functional status | one month, three months, six months, and twelve months after discharge
  Categorized as independent or not independent, based on ability to perform 6 activities of daily living (ADLs) and ability to walk.
Immune cell function | 1 week
  cytokine levels

CONTACTS AND LOCATIONS:
Overall Officials: John P Kress, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided